CLINICAL TRIAL: NCT01114308
Title: A Randomized, Placebo and Active-Controlled, Multi-Center Study of Probuphine in Patients With Opioid Dependence
Brief Title: A Six-Month Randomized Controlled Trial (RCT) of Probuphine Safety and Efficacy in Opioid Addiction
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Titan Pharmaceuticals (Industry)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PRO-806; 1RC2DA028910-01 (NIH)
Record Dates: First submitted 2010-04-27; First posted 2010-05-03 (Estimated); Last update posted 2018-12-31 (Actual); Status verified 2017-06

CONDITIONS: Opioid Dependency
Keywords: opioid dependence; opioid addiction; buprenorphine; implant; methadone; heroin; suboxone; opioid pain medication; opioid withdrawal
MeSH Terms: conditions — Opioid-Related Disorders | interventions — Buprenorphine; Buprenorphine, Naloxone Drug Combination

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Probuphine (Experimental): Patients are first inducted on SL BPN then switched to 4 buprenorphine implants
  Interventions: Drug: Probuphine (buprenorphine implant)
- placebo implant (Placebo Comparator): patients are first inducted on SL BPN then switched to 4 placebo implants
  Interventions: Drug: placebo implant
- sublingual buprenorphine (Active Comparator): patients are inducted on SL BPN, then continue on SL BPN
  Interventions: Drug: Buprenorphine

INTERVENTIONS:
Drug: Probuphine (buprenorphine implant) — Implantable formulation of buprenorphine made of buprenorphine HCl/ethylene vinyl acetate, considered a drug.
  Arms: Probuphine
Drug: placebo implant — Implant contains ethylene vinyl acetate
  Arms: placebo implant
Drug: Buprenorphine — sublingual buprenorphine/naloxone tablets
  Other Names: Suboxone
  Arms: sublingual buprenorphine

SUMMARY:
Probuphine (buprenorphine implant) is an implant placed just below the skin containing buprenorphine (BPN). BPN is an approved treatment for opioid dependence. This study will confirm the efficacy of Probuphine vs. placebo and compare Probuphine treatment verses treatment with sublingual buprenorphine in the treatment of patients with opioid dependence.

ELIGIBILITY:
Inclusion Criteria:

* Voluntarily provide written informed consent prior to the conduct of any study-related procedures
* Male or female, 18-65 years of age
* Meet DSM-IV-TR criteria for current opioid dependence
* Females of childbearing potential or a fertile male, must use a reliable means of contraception

Exclusion Criteria:

* Current diagnosis of Acquired Immune Deficiency Syndrome (AIDS)
* Received any medication-assisted treatment for opioid dependence (e.g., methadone, BPN) within the previous 90 days
* Current diagnosis of chronic pain requiring opioids for treatment
* Candidates for short-term opioid treatment (<6 months) only, or opioid detoxification therapy
* Pregnant or lactating female?
* Previous hypersensitivity or allergy to BPN, EVA-containing substances, or naloxone
* Current use of agents metabolized through Cytochrome P450 3A4 (CYP 3A4) such as azole antifungals (e.g., ketoconazole), macrolide antibiotics (e.g., erythromycin), or protease inhibitors (e.g., ritonavir, indinavir, and saquinavir)
* History of coagulopathy within the past 90 days, and/or current anti-coagulant therapy such as warfarin
* Meet the DSM-IV-TR criteria for dependence on any other psychoactive substances other than opioids or nicotine (e.g., alcohol, sedatives)
* Significant medical or psychiatric symptoms, cognitive impairment, or other factors which in the opinion of the Investigator would preclude compliance with the protocol, subject safety, adequate cooperation in the study, or obtaining informed consent
* Current medical conditions such as severe respiratory insufficiency that may prevent the subject from safely participating in study, or any pending legal action that could prohibit participation or compliance in the study
* Exposure to any investigational drug within the previous 8 weeks
* Previous exposure to Probuphine, or prior implantation with a placebo implant in the context of a Probuphine clinical trial
* Presence of aspartate aminotransferase (AST) levels greater than or equal to 3 X the upper limit of normal, alanine aminotransferase (ALT) levels greater than or equal to 3 X the upper limit of normal, total bilirubin greater than or equal to 1.5 X the upper limit of normal, or creatinine greater than 1.5 X upper limit of normal on the screening laboratory assessments
* Clinically significant low platelet count on the screening laboratory assessments

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 287 (Actual)
Dates: Start 2010-04; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
CDF of the percent of urine samples negative for opioids in Probuphine and Placebo groups from weeks 1-24 | 1-24 weeks
CDF of the percent of urine samples negative for opioids from weeks 1-24 with imputation based on illicit drug use self-report data for Probuphine and placebo groups | 1-24 weeks

SECONDARY OUTCOMES:
CDF of the percent of urine samples negative for opioids from weeks 1-16 | 1-16 weeks
CDF of the percent of urine samples negative for opioids from weeks 17-24 | 17-24 weeks
Difference of proportion of urine samples negative for illicit opioids over 24 weeks of treatment for Probuphine vs. SL BPN | 24 weeks

OTHER OUTCOMES:
Percent urines negative for illicit opioids | 24 weeks
Percent of study completers | 24 weeks
Mean total score on the SOWS | 24 weeks
Mean total score on the COWS | 24 weeks
Mean subjective opioid craving assessment using Visual Analog Scale (VAS) | 24 weeks
Patient-rated Clinical Global Improvement (CGI) | 24 weeks
Physician-rated Clinical Global Improvement (CGI) | 24 weeks
Mean total number of weeks of abstinence | 24 weeks
Mean maximum period of continuous abstinence | 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Katherine L. Beebe, Ph.D., Principal Investigator — Titan Pharmaceuticals
Locations (20):
- United States (20):
  - David Geffen School of Medicine at UCLA, Los Angeles, California
  - Synergy Clinical Research Center, National City, California
  - North County Clinical Research, Oceanside, California
  - Friends Research Institute, Torrance, California
  - Amit Vijapura, MD, Jacksonville, Florida
  - Operation PAR, Inc. - TC Campus, Largo, Florida
  - Fidelity Clinical Research, Inc., Lauderhill, Florida
  - Scientific Clinical Research, Inc., North Miami, Florida
  - BPRU, Behavioral Biology Research Center, Baltimore, Maryland
  - SSTAR: Stanley Street Treatment and Resources, Inc., Fall River, Massachusetts
  - Precise Research Centers, Flowood, Mississippi
  - PsychCare Consultants Research, St Louis, Missouri
  - New York VA Medical Center, NYU School of Medicine, New York, New York
  - St. Luke's Roosevelt Hospital Center, New York, New York
  - Duke University, Duke Addictions Program, Durham, North Carolina
  - University of Cincinnati, Cincinnati, Ohio
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Carolina Clinical Trials, Inc., Charleston, South Carolina
  - University of Vermont, Burlington, Vermont
  - Providence Behavioral Health Services, Everett, Washington

REFERENCES:
- [Derived] Rosenthal RN, Ling W, Casadonte P, Vocci F, Bailey GL, Kampman K, Patkar A, Chavoustie S, Blasey C, Sigmon S, Beebe KL. Buprenorphine implants for treatment of opioid dependence: randomized comparison to placebo and sublingual buprenorphine/naloxone. Addiction. 2013 Dec;108(12):2141-9. doi: 10.1111/add.12315. Epub 2013 Sep 18. PMID 23919595
- See also: Related Info — http://www.titanpharm.com